CLINICAL TRIAL: NCT07102459
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study Evaluating the Efficacy and Safety of LTG-001 for Acute Pain After an Abdominoplasty
Brief Title: An Efficacy and Safety Study of LTG-001 Following Abdominoplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Latigo Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LTG-001-010
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-07

CONDITIONS: Acute Pain; Postoperative Pain Control
Keywords: Acute Pain; Abdominoplasty
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LTG-001 High Dose (Experimental): High Dose LTG-001
  Interventions: Drug: Experimental: LTG-001 High Dose
- LTG-001 Low Dose (Experimental)
  Interventions: Drug: Experimental: LTG-001 Low Dose
- HB/APAP (Active Comparator)
  Interventions: Drug: Active Comparator: HB/APAP
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Experimental: LTG-001 High Dose — High Dose Active
  Arms: LTG-001 High Dose
Drug: Experimental: LTG-001 Low Dose — Lower Dose Active
  Arms: LTG-001 Low Dose
Drug: Active Comparator: HB/APAP — Active Comparator
  Arms: HB/APAP
Drug: Placebo Comparator — Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if LTG-001 works to treat post-operative / acute pain after an abdominoplasty procedure. It will also learn more information on the safety of LTG-001.

The main questions it aims to answer are:

Does drug LTG-001 treat the acute pain after surgical abdominoplasty over 48 hours? How tolerable is LTG-001 over 48 hours? What dose of LTG-001 is better for treating post-operative / acute pain?

Participants will:

Take LTG-001 bid after the surgical abdominoplasty. Remain at the clinic for approximately 48 hours during study dosing and return after two weeks for a safety check up. Report the pain relief during the 48 hours to record changes in the post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female aged 18 to 50 years
* Scheduled to undergo an elective "partial" abdominoplasty under general anesthesia
* Has a body BMI 18.0 to 35 kg/m2
* Has signed informed consent and will comply with the requirements and restrictions of the study
* Meet lifestyle, medication, or other study restrictions
* Subject must agree to study required use of birth control
* Post-surgical (abdominoplasty) pain must meet the study threshold

Exclusion Criteria:

* Inability to take oral medications
* Prior abdominoplasty or a prior intra-abdominal and/or pelvic surgery (including hysterectomy and Cesarean section) that resulted in any complications
* History of impaired hepatic function or heart disease.
* Abnormal liver laboratories or other lab abnormality indicative of serious medical condition
* Sensory abnormality that would confound post-surgery pain assessments
* Chronic use of NSAIDs, benzodiazepines, opioid use within the last year, use of medications that prolong QTc intervals, or other dietary and medication restrictions
* A subject with sleep apnea and/or on a home continuous positive airway pressure machine.
* Positive drug screen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
SPIDr0-48 | 48 hours
  Time-weighted SPIDr0-48 after the first dose of study drug.

SECONDARY OUTCOMES:
Total Opioid Rescue | 48 hours
  Total opioid rescue medication consumption from 0 48 hours, using MMEs
No Opioid requirement | 48 hours
  Proportion of participants requiring no opioid rescue medication over 48 hours
Nausea and Vomiting | 48 hours
  Incidence of nausea or vomiting
2-Point NPRS Reduction | 48 hours
  Time to ≥2-point reduction in NPRS from baseline
1-Point NPRS Reduction | 48 Hours
  Time to ≥1-point reduction in NPRS from baseline
PID at 60 minutes | 1 hour
  Time-specific PID at 60 minutes
SPID r0-24 | 24 hours
  Time-weighted SPIDr0-24 after the first dose of study drug
Patient Global Assessment | 48 Hours
  Proportion of participants with favorable PGA of study drug at end of treatment

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Arizona Research Center, Phoenix, Arizona
  - CenExel ACMR, Atlanta, Georgia
  - HD Research LLC, Houston, Texas
  - Endeavor Clinical Research, San Antonio, Texas
  - JBR Clinical Research (CenExel), Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No